CLINICAL TRIAL: NCT07196332
Title: Recovering Sleep After Trauma
Acronym: REST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Heart and Armor Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25-1574
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Trauma and Stressor Related Disorders; Mental Disorders; Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic; Motor Vehicle Collision
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Mental Disorders; Stress Disorders, Traumatic | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Behavioral Treatment for Insomnia (BBTI) (Experimental): Four sessions of telehealth-delivered brief behavioral treatment for insomnia
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia (BBTI)
- Progressive Muscle Relaxation Training (PMRT) (Active Comparator): Four sessions of telehealth-delivered progressive muscle relaxation training
  Interventions: Behavioral: Progressive Muscle Relaxation Training (PMRT)

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia (BBTI) — In the first week, treatment consists of a 60-minute video individual intervention session; in the second week, participants receive a 30-minute phone call; in the third week, treatment consists of a 45-minute video individual session; the final session consists of a 30-minute phone call. BBTI emphasizes behavioral elements of insomnia treatment. Treatment begins with sleep education and discussion of homeostatic and circadian mechanisms of human sleep regulation. Next, a series of interventions are employed that are derived from sleep restriction and stimulus control techniques.
  Arms: Brief Behavioral Treatment for Insomnia (BBTI)
Behavioral: Progressive Muscle Relaxation Training (PMRT) — In the first week, treatment consists of a 60-minute video individual intervention session; in the second week, participants receive a 30-minute phone call; in the third week, treatment consists of a 45-minute video individual session; the final session consists of a 30-minute phone call. Treatment begins with learning how to alternately tense and relax 14 major muscle groups, and then to use progressively more efficient tensing-relaxing and passive relaxation exercises, with sessions used to teach techniques and problem-solve barriers to its daily use.
  Arms: Progressive Muscle Relaxation Training (PMRT)

SUMMARY:
The main objective of this pilot trial is to assess the feasibility and preliminary efficacy of telehealth-delivered behavioral therapy to reduce the development of posttraumatic stress and depressive symptoms following motor vehicle collision among individuals at high risk. This pilot trial will provide the data necessary to design and support a large-scale trial.

DETAILED DESCRIPTION:
Each year, more than 40 million Americans present to US emergency departments (EDs) for evaluation after traumatic stress exposure. The overwhelming majority of these individuals are discharged home after evaluation. A wealth of data demonstrates that the development of adverse posttraumatic neuropsychiatric sequelae such as posttraumatic stress disorder (PTSD) is common in this population, and that individuals with a history of traumatic stress exposure and/or posttraumatic stress symptoms-such as military veterans-are at increased risk. Unfortunately, no secondary preventive interventions are currently widely available that can prevent PTSD among those at high risk. This pilot REST trial will assess the ability of brief behavioral treatment for insomnia (BBTI) to reduce the incidence and severity of PTSD and depression after one of the most common traumatic stress exposures in industrialized countries, motor vehicle collision (MVC). BBTI is an evidence-based, low-cost intervention that has been demonstrated to be effective in treating insomnia and reducing PTSD symptoms. However, BBTI has never been tested as a secondary preventive intervention for PTSD and depression. In addition, the efficacy of BBTI when administered as a telehealth intervention has never been assessed. This REST pilot trial will randomize 20 (N=20) individuals who present to a study ED for care after MVC to four sessions of brief behavioral treatment for insomnia (BBTI) versus a progressive muscle relaxation training (PMRT) control. Both interventions will be administered via telehealth, with 10 individuals receiving BBTI and 10 receiving PMRT. Each therapist will administer both interventions. Participants will be assessed via traditional self-report surveys and sleep diaries. Results of this trial will demonstrate the feasibility and potential efficacy of BBTI to prevent the development of PTSD and depression after traumatic stress exposure and will provide the data necessary to design/support a large-scale trial. Developing preventive interventions to reduce PTSD and depression among individuals experiencing civilian trauma exposures would reduce suffering and considerable costs associated with these disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Alert and oriented at time of screening
2. Written and spoken English
3. Age 18-65
4. Presents to the ED within 72 hours of MVC
5. Discharged home after ED evaluation
6. Has an email and mailing address
7. Owns a smartphone compatible with iOS or Android, has not experienced service interruption due to non-payment in the past year, and has maintained the same phone number for at least one year
8. Meets PTSD risk score criteria (score of ≥ 16 on the PTSD risk stratification tool)
9. Willing to participate in four remote therapy sessions

Exclusion Criteria:

1. Age <18 or >65
2. Pregnant
3. Prisoner or in police custody
4. Present to ED >72 hours after trauma
5. Admitted to the hospital after ED evaluation
6. Severely injured (e.g., severely broken bones) as a result of the MVC that, in the opinion of the investigator, may impact PTSD trajectories
7. Had a change in psychiatric medication or psychotherapy regimen within 1 month of enrollment
8. Currently receiving or planning to receive evidence-based treatments that directly target insomnia or PTSD (e.g., CBT-I, Cognitive Processing Therapy, or Prolonged Exposure Therapy)
9. MVC was self-inflicted or occupation-related
10. Report or indicate that they are experiencing ongoing domestic violence
11. Has conditions that may be associated with comorbid insomnia, including a lifetime history of any psychiatric disorder with psychotic features, manic or hypomanic episodes. We will not exclude individuals based on any other mental health condition, including depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes in PTSD Symptom Severity Over Time | Baseline, Week 4, Week 8, Month 3
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure designed to assess PTSD symptoms as defined by the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5). The PCL-5 will be completed in reference to the motor vehicle collision (MVC) that occurred just before enrollment into the study. Each item of the PCL-5 is scored on a five-point scale ranging from 0 ("not at all") to 4 ("extremely"). Items are summed to provide a total severity score (range = 0-80), with higher scores indicating greater symptom severity. PTSD symptom severity will be compared between treatment groups over time.
Recruitment Rates | Baseline
  To assess the feasibility of the study recruitment protocol, the proportion of eligible participants who enroll in the study and are randomized will be calculated.
Retention Rates | Month 3
  To assess feasibility of the study protocol, the proportion of participants who complete the study protocol, according to study arm and in total, will be calculated.
Treatment Completion Rates | Week 4
  To assess feasibility of the treatment protocol, treatment completion rates will be calculated according to the study arm and in total. Treatment completers will be defined as participants who complete at least 3 out of 4 REST or control sessions.

SECONDARY OUTCOMES:
Change in Depressive Symptom Score Over Time | Baseline, Week 4, Week 8, Month 3
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form 8b is an 8-item scale developed to assess depression in individuals 18 and older. Each item is rated on a five-point scale. For this study, response options are slightly altered for greater consistency across measures and precision in response levels (i.e., 1 = "never" is changed to none of the time and 5 = "always" is changed to "all or almost all of the time."). Items are summed to provide a total severity score (range = 8-40), with higher scores indicating greater severity of depression. Depressive symptom severity will be compared between treatment groups over time.
Change in Somatic Score Symptoms Over Time | Baseline, Week 4, Week 8, Month 3
  Somatic symptoms will be assessed using a modified version of the Pennebaker Inventory of Limbic Languidness (PILL), which assesses the frequency of common physical symptoms and sensations. Each item is scored on a 0-10 scale where 0 indicates no problems. Number of moderate to severe somatic symptoms (scores ≥ 4) will be compared between groups.
Change in Pain Symptom Severity and Extent Over Time | Baseline, Week 4, Week 8, Month 3
  Pain severity and extent will be evaluated using a modified version of the Regional Pain Scale, where each item is scored on a 0-10 numeric rating with 0 indicating no pain and 10 indicating severe pain. Pain symptom severity and extent will be compared between treatment groups over time.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel McLean, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared on request provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Time Frame: Beginning 12 months following publication and continuing for 36 months.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.